CLINICAL TRIAL: NCT06190678
Title: An Open-label, Nonrandomized, Single-dose, Parallel-group, Safety, Tolerance, and Pharmacokinetic Study of LOXO-305 Administered to Fasted Renally Impaired Male and Female Subjects and Fasted Matched-control Healthy Subjects
Brief Title: Study of Pirtobrutinib (LOXO-305) in Participants With Impaired Kidney Function and Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-BTK-20013; J2N-OX-JZNG (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pirtobrutinib (Normal Renal Function) (Experimental): Participants with normal renal function (eGFR >= 90 mL/min/1.73 m2) received a single dose of Pirtobrutinib 200 milligrams (mg) administered orally on Day 1.
  Interventions: Drug: Pirtobrutinib
- Pirtobrutinib (Severe Renal Impairment) (Experimental): Participants with severe renal impairment (eGFR: < 30 mL/min/1.73 m2) received a single dose of Pirtobrutinib 200 mg administered orally on Day 1.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally
  Other Names: LOXO-305, LY3527727

SUMMARY:
The main purpose of this study is to measure how much of pirtobrutinib (LOXO-305) gets into the bloodstream and how long it takes the body to eliminate it in participants with impaired kidney function and healthy participants. The side effects and tolerability of pirtobrutinib will also be evaluated. Participation could last around 46 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants with impaired renal function [estimated Glomerular Filtration Rate (eGFR): < 90 milliliters per minute (mL/min) per 1.73 square meters (m2)] and healthy participants with normal renal function [(eGFR: ≥ 90 mL/min/1.73 m2)].
* Males and females of non-childbearing potential.
* Within body mass index (BMI) range 18.5 to 40.0 kilograms per square meter (kg/m²).
* Participants will be in good health, based on medical history, physical examination findings, vital signs, 12 lead electrocardiogram (ECG), or clinical laboratory tests, as determined by the Investigator (or designee).
* Able to comply with all study procedures, including the 8-night stay at the Clinical Research Unit and follow-up phone call.

Exclusion Criteria:

* History or presence of any of the following, deemed clinically significant by the Investigator (or designee), and/or Sponsor:

  1. liver disease
  2. pancreatitis
  3. peptic ulcer disease
  4. intestinal malabsorption
  5. gastric reduction surgery
  6. history or presence of clinically significant cardiovascular disease.
* Participants with out-of-range, at-rest vital signs.
* Abnormal laboratory values determined to be clinically significant by the Investigator (or designee).
* Clinically significant abnormality, as determined by the Investigator (or designee), from physical examination.
* Participation in any other investigational study drug trial involving administration of any investigational drug in the past 30 days or 5 half-lives, whichever was longer, prior to the first dose administration (Day 1).
* Use or intention to use any prescription or over-the-counter medications within 14 days prior to the first dose administration (Day 1) and through end of trial.
* History or presence, upon clinical evaluation, of any illness that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results, or put the participant at undue risk.
* Donation of blood from 56 days prior to Screening, plasma or platelets from 4 weeks prior to Screening.
* Receipt of blood products within 2 months prior to Check-in (Day -1).
* Significant history of hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renée Ward, MD, PhD, Study Director — Loxo Oncology
Locations (5):
- United States (5):
  - Orange County Research Institute, Anaheim, California
  - Riverside Clinical Research, Edgewater, Florida
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Prism Research, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with normal renal function, as well as those with mild, moderate, or severe renal impairment, were initially planned to be enrolled in the study. However, based on the results of the interim analysis, it was decided that including participants with mild or moderate renal impairment was not required.
Groups:
- Pirtobrutinib (Normal Renal Function): Participants with normal renal function (eGFR: >= 90 mL/min/1.73 m2) received a single dose of Pirtobrutinib 200 mg administered orally on Day 1.
Period: Overall Study
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Started | 8 | 8
Received Dose of Pirtobrutinib | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (4.06) | 64 (6.93) | 61.1 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Pirtobrutinib
Description: PK: Cmax of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: All participants who received a dose of Pirtobrutinib, had at least 1 quantifiable plasma concentration of Pirtobrutinib and had at least 1 PK parameter computed. Subjects were excluded from the analysis if they experienced an AE of vomiting that occurred at or before 2 times the median Tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
nanogram per milliliter (ng/mL) | 3450 (19.7) | 2910 (30.9)

2. Primary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of Pirtobrutinib
Description: PK: Tmax of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
hours | 3 [1.50 to 8] | 2 [0.75 to 3]

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) of Pirtobrutinib
Description: PK: AUC0-t of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
hour*nanogram per milliliter (h*ng/mL) | 73800 (18.6) | 103000 (34.2)

4. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) of Pirtobrutinib
Description: PK: AUC0-inf of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
hour*nanogram per milliliter (h*ng/mL) | 75100 (18.3) | 107000 (35.3)

5. Primary Outcome: PK: Percentage Extrapolation for AUC0-inf (%AUCextrap) of Pirtobrutinib
Description: PK: %AUCextrap of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUCextrap
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
percentage of AUCextrap | 1.55 (46.2) | 4.05 (28.3)

6. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (λZ) of Pirtobrutinib
Description: PK: λZ of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour (1/h)
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
1/hour (1/h) | 0.0317 (22.6) | 0.0183 (10.8)

7. Primary Outcome: PK: Apparent Plasma Terminal Elimination Half-life (t½) of Pirtobrutinib
Description: PK: t½ of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
hours | 21.9 (22.6) | 37.8 (10.8)

8. Primary Outcome: PK: Apparent Systemic Clearance (CL/F) of Pirtobrutinib
Description: PK: CL/F of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
liter per hour (L/h) | 2.66 (18.3) | 1.86 (35.3)

9. Primary Outcome: PK: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of Pirtobrutinib
Description: PK: Vz/F of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
Liter (L) | 84 (19.2) | 102 (29.4)

10. Primary Outcome: PK: Mean Residence Time (MRT) of Pirtobrutinib
Description: MRT is the average time a drug molecule stays in the body, calculated from the AUC0-inf.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
hours | 27.6 (13.3) | 48.8 (10.4)

11. Primary Outcome: PK: Unbound Cmax (Cmax,u) of Pirtobrutinib
Description: Cmax,u was calculated by multiplying Cmax by Fu (i.e., Cmax*Fu).
  Fu represents the unbound fraction, which is the portion of the drug in the bloodstream that is unbound to plasma proteins. It is expressed as a decimal and will be calculated from protein binding concentration data as the unbound drug concentration divided by the total drug concentration in plasma. The concentrations of total and unbound drug were determined in a sample of predose plasma fortified with a known concentration of drug.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
nanogram per milliliter (ng/mL) | 131 (25.5) | 110 (26.6)

12. Primary Outcome: PK: Unbound AUC0-t (AUC0-t,u) of Pirtobrutinib
Description: AUC0-t,u was calculated by multiplying AUC0-t by Fu (i.e., AUC0-t*Fu).
  Fu represents the unbound fraction, which is the portion of the drug in the bloodstream that is unbound to plasma proteins. It is expressed as a decimal and will be calculated from protein binding concentration data as the unbound drug concentration divided by the total drug concentration in plasma. The concentrations of total and unbound drug were determined in a sample of predose plasma fortified with a known concentration of drug.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
hour*nanogram per milliliter (h*ng/mL) | 2800 (24.7) | 3870 (36.6)

13. Primary Outcome: PK: Unbound AUC0-inf (AUC0-inf,u) of Pirtobrutinib
Description: AUC0-inf,u was calculated by multiplying AUC0-inf by Fu (i.e., AUC0-inf*Fu).
  Fu represents the unbound fraction, which is the portion of the drug in the bloodstream that is unbound to plasma proteins. It is expressed as a decimal and will be calculated from protein binding concentration data as the unbound drug concentration divided by the total drug concentration in plasma. The concentrations of total and unbound drug were determined in a sample of predose plasma fortified with a known concentration of drug.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
hour*nanogram per milliliter (h*ng/mL) | 2850 (24.8) | 4040 (37.4)

14. Primary Outcome: PK: Unbound CL/F (CL/F,u) of Pirtobrutinib
Description: CL/F,u was calculated by multiplying CL/F by Fu (i.e., CL/F*Fu).
  Fu represents the unbound fraction, which is the portion of the drug in the bloodstream that is unbound to plasma proteins. It is expressed as a decimal and will be calculated from protein binding concentration data as the unbound drug concentration divided by the total drug concentration in plasma. The concentrations of total and unbound drug were determined in a sample of predose plasma fortified with a known concentration of drug.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
liter per hour (L/h) | 70.2 (24.8) | 49.5 (37.4)

15. Primary Outcome: PK: Unbound Vz/F (Vz/F,u) of Pirtobrutinib
Description: Vz/F,u was calculated by multiplying Vz/F by Fu (i.e., Vz/F*Fu).
  Fu represents the unbound fraction, which is the portion of the drug in the bloodstream that is unbound to plasma proteins. It is expressed as a decimal and will be calculated from protein binding concentration data as the unbound drug concentration divided by the total drug concentration in plasma. The concentrations of total and unbound drug were determined in a sample of predose plasma fortified with a known concentration of drug.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
Number analyzed (Participants) | 8 | 7
Liter (L) | 2210 (16.8) | 2700 (35.2)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To Day 17)
Description: All participants who received a dose of Pirtobrutinib.
Arm/Group | Pirtobrutinib (Normal Renal Function) | Pirtobrutinib (Severe Renal Impairment)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pirtobrutinib (Normal Renal Function) (N=8) | Pirtobrutinib (Severe Renal Impairment) (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT06190678/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT06190678/SAP_001.pdf